CLINICAL TRIAL: NCT05104879
Title: The Patient's Experience With Physician Assistant Providers: a Descriptive Survey and Randomized Intervention
Brief Title: The Patient's Experience With Physician Assistant Providers (PEPAP)
Acronym: PEPAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Desert Orthopedic Center (Other)
Responsible Party: Principal Investigator, Russell Nevins, M.D., Orthopaedic Surgeon, Desert Orthopedic Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: DOC0001
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Joint Diseases, Midlevel Providers, Nurse Practitioners, Physician Assistants, Patient Perceptions, Patient Preferences
MeSH Terms: conditions — Joint Diseases; Patient Preference

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biosketch Card (Experimental): Patients within the experimental group received a biosketch card during rooming, pre-clinician encounter, and were not informed about their involvement. To blind the outcome measure, the research assistant did not explain the reason for the card upon rooming the patient nor did they inform the midlevel provider.
  Interventions: Other: Biosketch Card
- No Card (No Intervention): No bio sketch card was provided to these participants.

INTERVENTIONS:
Other: Biosketch Card — The experimental group received a biosketch card during rooming, pre-clinician encounter that gave an overview of the midlevel providers qualifications.
  Arms: Biosketch Card

SUMMARY:
Our investigation was a prospective cross-sectional survey evaluating the patient experience to new patients that presented to an outpatient private practice specialized in total joint reconstruction. New patients seeing a PA during their initial visit were randomized to intervention and control groups and all were given a descriptive survey at checkout. Inclusion criteria (1) new patient (2) English speaking (3) appointment with PA. There was no exclusion criteria. Eligible patients were randomized to the intervention group (received biosketch card) or the control group (no card) using random number generator. Patients within the intervention group received a biosketch card during rooming, pre-clinician encounter, and were not informed about involvement. Both groups received standard care that was independent of the study. To blind the outcome measure, the research assistant did not explain the reason for the card upon rooming. The provider PA was not informed which patient received the card. Upon discharge, the patient completed a five-question survey regarding the clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* New Patient
* Appointment with a PA

Exclusion Criteria:

* Non-English Speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Survey | Immediately following the visit
  Five question survey following the visit

IPD SHARING:
Plan to Share IPD: No
We won't be sharing any of the individual participant data.